CLINICAL TRIAL: NCT06698536
Title: OBPM_COYOTE2024 Physiological Data Recording With the Calibration-free Optical Aktiia G2C Device at Fingertip and Wrist, Alongside the Aktiia Oscillometric Cuff: a Single-center, Prospective Clinical Study
Brief Title: OBPM_COYOTE2024 Physiological Data Recording With the Calibration-free Optical Aktiia G2C Device at Fingertip and Wrist, Alongside the Aktiia Oscillometric Cuff
Acronym: COYOTE2024
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OBPM_COYOTE2024
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Study subjects are asked to stay seated while 3 successive measurements are taken with the device under investigation (BP and PR) and two references (Aktiia Bracelet G2 and Aktiia Init I1 oscillometric cuff).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aktiia G2C cohort (Other): Study subjects are asked to stay seated while 3 successive measurements are taken with the Aktiia G2C device under investigation (BP and PR) and two references (Aktiia Bracelet G2 and Aktiia Init I1 oscillometric cuff).
  Interventions: Device: Aktiia G2C

INTERVENTIONS:
Device: Aktiia G2C — Study subjects are asked to stay seated while 3 successive measurements are taken with the Aktiia G2C device under investigation (BP and PR) and two references (Aktiia Bracelet G2 and Aktiia Init I1 oscillometric cuff).

SUMMARY:
The present study, OBPM_COYOTE2024, with N = 255 participants minimum over 1 visit (lasting ~15min), has been designed to collect raw optical data with Aktiia.product-G2C Clinical investigational device together with Aktiia G2 Bracelet and Aktiia Init I1 oscillometric cuff within a cohort of subjects characterized by a wide variety of phenotypes. The resulting dataset will support research and development activities conducted by AKTIIA SA out of the study context.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 21 to 85yo
* Subjects or witnesses fluent in written and spoken French
* Subjects agreeing to attend the study visit and follow study procedures
* Subjects that have signed the informed consent form.

Exclusion Criteria:

* Amputated index fingers
* Damaged/injured skin at index fingers
* Damaged/injured skin at wrists
* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with diabetes
* Subjects with marked renal dysfunctions (eGFR < 30mL/min/1.73 m2)
* Subjects with untreated hyper-/hypothyroidism
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with an arteriovenous fistula
* Women in known pregnancy
* History of polyneuropathy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Data set build | Baseline
  Number of subjects including three assessments of blood pressure using Aktiia G2C Clinical, alongside three assessments of blood pressure with Aktiia Bracelet G2 and three values of blood pressure generated with the Aktiia Init I1 oscillometric cuff

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV Service de Néphrologie et d'Hypertension, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No